CLINICAL TRIAL: NCT05438277
Title: Incidence of Flare Reaction Following Shoulder Steroid Injections: Comparison of Depo-medrol (Methylprednisolone) and Kenalog (Triamcinolone)
Brief Title: Pain Increases After Shoulder Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Tyler J. Brolin, Principal Investigator, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 7001-XP
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Methylprednisolone; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- methylprednisolone acetate (MPA) (Experimental): subacromial or glenohumeral shoulder injection
  Interventions: Drug: Methylprednisolone (MPA)
- triamcinolone acetonide (TA) (Active Comparator): subacromial or glenohumeral shoulder injection
  Interventions: Drug: Triamcinolone Acetonide (TA)

INTERVENTIONS:
Drug: Methylprednisolone (MPA) — injection into subacromial or glenohumeral space with MPA
  Other Names: depomedrol
  Arms: methylprednisolone acetate (MPA)
Drug: Triamcinolone Acetonide (TA) — injection into subacromial or glenohumeral space with TA
  Other Names: kenalog
  Arms: triamcinolone acetonide (TA)

SUMMARY:
Compare FLARE reactions (increase in VAS by two or more points) in the first 48 hours following a shoulder injection.

DETAILED DESCRIPTION:
Corticosteroid injections are used to reduce pain and inflammation for various shoulder pathologies. Corticosteroid flare reaction is a well-described phenomenon that, despite being self-limited, causes significant pain and dysfunction. A flare reaction is defined for the purposes the study to be an increase of two or more points on a visual analog scale reported by the subject. Currently, there is a paucity of literature to drive the decision-making process between different corticosteroid medications. This study will compare the incidences of steroid flare reaction and three-month efficacy following methylprednisolone acetate (MPA) and triamcinolone acetonide (TA) corticosteroid injections into the glenohumeral joint or subacromial space.

Physicians administering a steroid injection in the shoulder will utilize MPA until 200 subjects have agreed to participate in this treatment arm. Enrollment will then be offered to 200 subjects utilizing TA for the shoulder injection. Subjects receive treatment for their shoulder pain regardless of willingness to participate in the follow up reported pain scores. There are no costs to subjects for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial or glenohumeral shoulder pain to be treated with steroid injection
* Fluent in written and oral English
* Willing and able to provide written consent
* Willing to complete follow up pain scores (visual analog score)

Exclusion Criteria:

* Unable to provide written consent
* Chronic pain syndrome
* Unwilling to complete follow up pain scores (visual analog score)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Brolin, MD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 421 patients were enrolled in the study. Out of these 421, 15 patients received bilateral shoulder injections. Thus, there were 436 total shoulders injected. The term used in the study to refer to the number of shoulders injected, rather than the number of patients, is "person-visits."
Units Other Than Participants: Person-visits
Period: Overall Study
Arm/Group | Methylprednisolone Acetate (MPA) | Triamcinolone Acetonide (TA)
Started | 205; 209 Person-visits (4 patients received bilateral shoulder injections) | 216; 227 Person-visits (11 patients received bilateral shoulder injections)
Completed | 205; 209 Person-visits | 216; 227 Person-visits
Not Completed | 0; 0 Person-visits | 0; 0 Person-visits

BASELINE CHARACTERISTICS:
Population: 4 patients in the MPA group received bilateral injections, for a total of 209 shoulders receiving a MPA injection. 11 patients in the TA group received bilateral injections, for a total of 227 shoulders receiving a TA injection. The name used in the study for the total number of injections, including bilateral injections, was "person-visits."
Units Other Than Participants: Person-visits
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone Acetate (MPA) | Triamcinolone Acetonide (TA) | Total
Number analyzed (Participants) | 205 | 216 | 421
Number analyzed (Person-visits) | 209 | 227 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.19 (13.54) | 60.64 (12.48) | 62.37 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 117 | 222
  Male | 100 | 99 | 199
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White American | 149 | 161 | 310
  African American | 52 | 50 | 102
  Others | 4 | 5 | 9
Injury/Pain Type [Count of Participants; unit: Participants]
  Acute | 105 | 90 | 195
  Chronic | 100 | 126 | 226

OUTCOME MEASURES:

1. Primary Outcome: Incidence of a Flare Reaction
Description: A flare reaction was defined as an increase of two or more points of Visual Analog Score (VAS) score during the first week following injection. The VAS is a patient reported pain score from zero to ten where zero is no pain and ten is the most pain.
Time Frame: Post-injection day 1 through 7
Population: The "Overall Number of Participants Analyzed" here reflects the number of person-visits for which data was able to be acquired. 16 person-visits in the MPA cohort were lost to follow-up during this time point, while 28 person-visits in the TA cohort were lost to follow-up during this time point. Loss to follow-up primarily was due to failure by subjects to mail their "home diary" VAS log.
Measure: Count of Units; unit: Person-visits
Units Other Than Participants: Person-visits
Arm/Group | Methylprednisolone Acetate (MPA) | Triamcinolone Acetonide (TA)
Number analyzed (Participants) | 205 | 216
Number analyzed (Person-visits) | 209 | 227
Person-visits
  Flare reaction (Yes) | 44 | 8
  Flare reaction (No) | 149 | 191
  Unknown | 16 | 28

ADVERSE EVENTS:
Description: Deaths, serious adverse advents, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Methylprednisolone Acetate (MPA) | Triamcinolone Acetonide (TA)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT05438277/Prot_SAP_000.pdf